CLINICAL TRIAL: NCT04396431
Title: The Effect of Nurse Health Education and Follow-up Programme on Sun Protection
Brief Title: The Effect of Nurse Health Education and Follow-up Programme on Sun Protection Behaviors of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, özüm erkin, associate prof, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 433178
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Nurse's Role; Cancer
Keywords: nursing; Transtheoretical model; sun protection; self-efficacy; decisional balance; prevention
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2 (Other): The intervention group was offered a six-hour training program based on the transtheoretical model in order to promote sun protection behavior and to reinforce self-efficacy.
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — The intervention group was offered a six-hour training program based on the transtheoretical model in order to promote sun protection behavior and to reinforce self-efficacy. The program was prepared by the researchers in consideration of the SunSmart Program implemented in Australia, the SunWise School Program developed by the United States Environmental Protection Agency. The program included various educational tools such as a sun protection story, activity book, PowerPoint presentations, cartoons, and puzzles.
  Refresher training was conducted 15 days, 1 month, and 2 months after the initial training. Sun protection behavior and self-efficacy of the children were evaluated at the beginning of the study and six months after the program. As gifts to support their sun protection behavior, the children were given an FDA-approved sunscreen with 50+ SPF, a white cotton short-sleeved T-shirt as protective clothing, sunglasses with 100% UV protection, and a wide-brimmed hat.

SUMMARY:
The aim of the study is to determine the effect of nurse health education and follow up program on sun protection behaviors of children. The study as a randomized controlled group was implemented in February- October 2014 in Turkey. After obtaining the parents' and the children's written consent, data were collected through face-to-face interviews using, the instruments (stages of change, the decisional balance scale, child and parental sun protection behavior form, self-efficacy form) on sun protection based on the transtheoretical model.

DETAILED DESCRIPTION:
Approximately 25% of lifelong sun exposure is formed prior to the age of 18. A significant correlation between exposure to ultraviolet radiation in childhood and skin cancer in adulthood draws attention to the importance of sun protection behaviors to be applied in this period. School-age children are easily reachable to promote preventive health behaviors. The aim of the study is to determine the effect of nurse health education and follow up program on sun protection behaviors of children. The study as a randomized controlled group trial was implemented in February- October 2014. Purposive nonprobability sampling was used to select 25 schools in Izmir Karşıyaka district and research was conducted in two schools where attending the children coming from medium families. Risk assessment for skin cancer was performed by Fitzpatrick classification with 260 children before the study. Out of these children, 144 were found to be risky and were randomized to intervention (n = 40) and control (n = 40) groups according to their age, gender, and skin type. In the survey, the effect size was identified as 0.73 by a 5% error and 80% confidence. After obtaining the parents' and the children's written consent, data were collected through face-to-face interviews using, the instruments (stages of change, the decisional balance scale, child and parental sun protection behavior form, self-efficacy form) on sun protection based on the transtheoretical model. Turkish validity and reliability study of the scale was conducted by Aygün and Ergün (2013). The intervention group was trained about sun protection behaviors in six sessions. Each session lasted 45 minutes. Refresher training was organized on the 15th day, on 1st month 2nd month after the first session. At the beginning and at the end of the program, decisional balance and self-efficacy of children were evaluated. Data were analyzed by frequencies, regression, Wilcoxon signed-rank test, paired-samples t-test, independent samples t-test, Mann-Whitney U test, Friedman's test, and Chi-square test. Written consent was taken from children and their parents, schools, and the local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 9
* have the consent of a parent
* Fitzpatrick skin type between 1 and 3

Exclusion Criteria:

* Fitzpatrick skin type between 4 and 6

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — school-aged children
Enrollment: 80 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
self-efficacy | 6 months
  examines self efficacy regarding protection from the sun. It is also scored on a five-point scale (1 - not at all confident, 2 - not very confident, 3 - moderately confident, 4 - very confident, and 5 - extremely confident)

SECONDARY OUTCOMES:
sun protection behavior | 6 months
  measures the incidence of sun protection behavior when outdoors for periods longer than 15 minutes. It is scored on a five-point scale ranging from 1 to 5 (1 - never, 2 - rarely, 3 - sometimes, 4 - often, and 5 - always)

IPD SHARING:
Plan to Share IPD: No